CLINICAL TRIAL: NCT00844883
Title: Phase II Trial of Sorafenib Combined With Doxorubicin Eluting Bead-Transarterial Chemoembolization (LC Bead-TACE) for Patients With Hepatocellular Carcinoma
Brief Title: Study of Sorafenib and Transarterial Chemoembolization (TACE) to Treat Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Bayer (Industry); Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J08110
Record Dates: First submitted 2009-02-04; First posted 2009-02-16 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Hepatocellular Carcinoma; Hepatoma
Keywords: primary liver cancer; sorafenib; Nexavar; doxorubicin; drug eluting beads; transarterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib and drug eluting beads (Experimental): single arm
  Interventions: Drug: sorafenib; Procedure: LC Bead-TACE

INTERVENTIONS:
Drug: sorafenib — sorafenib: given 400 mg twice per day for as long as it is beneficial
  Other Names: sorafenib (Nexavar)
Procedure: LC Bead-TACE — LC Beads loaded with doxorubicin
  Doxorubicin loaded LC Beads: given intra-arterially into the liver, up to fours times in a 6 month period
  Other Names: LC Beads manufactured by Biocompatibles

SUMMARY:
This study will combine two therapies to treat patients with unresectable hepatocellular carcinoma; sorafenib, and drug eluting beads delivered intra-arterially. The purpose of the study is to establish the safety and the effectiveness of the combination therapy. The investigators hypothesize that the combination of the two therapies will not result in greater toxicities to patients than that expected for either therapy given alone.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable hepatocellular carcinoma (HCC) patients with liver-predominant disease as described in section 5.1, or patients with hepatocellular carcinoma who refuse surgery. No more than 30% of the cohort should have macrovascular invasion and/or asymptomatic extrahepatic disease. Multifocal HCC is acceptable, no diffuse HCC.
2. Age > 18 years old
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
4. Childs class of A or B (up to 7) (see Table 5.0)
5. Adequate end-organ function as manifested by:

   * Absolute neutrophil count of > 1500/mm3 and platelets > 50,000/mm3
   * Creatinine ≤ 2.0
   * Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) < 5 x upper limit of normal (ULN)
   * Total bilirubin of ≤ 3
   * Albumin > 2.0
   * International normalized ratio (INR) < 2.0
   * Leukocyte count >3000 cells/mm3
6. Amylase and lipase ≤ 1.5 the upper limit of normal
7. Patients who have received previous hepatic surgery , radiofrequency ablation (RFA), percutaneous ethanol injection (PEI), or cryoablation are eligible if target lesion(s) have not been treated and local therapy completed > 6 weeks prior to entry.
8. Left ventricular ejection fraction ≥ 45%
9. Patients with asymptomatic HIV infection are not eligible
10. Willingness of male and female subjects, who are not surgically sterile or post menopausal, to use reliable methods of birth control for the duration of the study and for 30 days after the last dose of study medication.
11. Patient must have signed informed consent prior to registration on study.
12. Resolution of all acute toxic effects of any prior local treatment to Common Terminology Criteria for Adverse Events (CTCEA) Grade 1 or 0.
13. At least one tumor lesion can be accurately measured in at least one dimension according to RECIST. The lesion has not been previously treated with local therapy (such as surgery, radiation therapy, RFA, PEI, or cryoablation) unless it has shown progression in the interim.

Exclusion Criteria:

1. Patients unable to swallow oral medications
2. Prior embolization, systemic or radiation therapy for HCC (liver)
3. Tumor burden in the liver exceeding 70%.
4. Complete occlusion of the entire portal venous system
5. Ascites refractory to diuretic therapy (minimal or trace on imaging is acceptable)
6. Previous or concurrent cancer that is distinct in primary site or histology from HCC, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis, and T1). Any cancer curatively treated > 3 years prior is permitted.
7. Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
8. History of bleeding within the past 4 weeks (unless deemed by PI as clinically insignificant, for ex., a brief episode of epistaxis)
9. Any contraindication to doxorubicin administration
10. Evidence of severe or uncontrolled systemic diseases,
11. Congestive cardiac failure > New York Heart Association (NYHA) class 2, myocardial ischemia within 6 months, active coronary artery disease, cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin, unstable angina, or laboratory finding that in the view of the investigator makes it undesirable for the patient to participate in the trial
12. Any prior history of hypertensive crisis or hypertensive encephalopathy
13. History of stroke or transient ischemic attack within 6 months prior to study enrollment
14. Inadequately controlled hypertension (defined as systolic blood pressure of 150/100 mmHg on antihypertensive medications) (patients with treated hypertension are eligible)
15. Significant vascular disease (e.g., aortic aneurysm, aortic dissection, peripheral vascular disease)
16. History of organ allograft
17. Presence of grade > 2 hepatic encephalopathy (see Appendix D)
18. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an additional experimental drug
19. Evidence of bleeding diathesis or coagulopathy or on warfarin. Note: If a patient has been on coumadin for a period of 1 month and has been stable, they may be accepted into the protocol.
20. Presence of clinically evident central nervous system or brain metastases
21. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, anticipation of need for major surgical procedure during the course of the study
22. Vascular anatomy that precludes catheter placement or injection of LC Bead microspheres
23. Presence of collateral vessel pathways potentially endangering normal territories during embolization
24. Pregnant (positive pregnancy test) or lactating
25. Inability to comply with study and/or follow-up procedures
26. Life expectancy of less than 12 weeks
27. Child B8, B9 and C
28. ECOG ≥ 2
29. Patients with concomitant HIV infection or AIDS-related or serious acute or chronic illness
30. Presence of porto-systemic shunt
31. Severe atheromatosis
32. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of study results
33. Active clinically serious infections (>grade 2)
34. Patients receiving therapy for hepatitis A, B, or C.
35. Patients with obvious and/or symptomatic extrahepatic disease. Findings of uncertain significance, such as lung lesions less than 10 mm in diameter or enlarged periportal lymph nodes will not exclude patients, however, findings highly suspicious for metastatic HCC will exclude patients from this study.
36. Any contraindication for an arterial procedure such as impaired clotting tests (platelet count < 50.000/mm3 or prothrombin activity < 50 percent)
37. Any contraindication for systemic chemotherapy administration (serum bilirubin > 3mg/dL, leukocyte count < 3.000 cells/mm3)
38. Any contraindication for sorafenib administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients diagnosed with unresectable hepatocellular carcinoma who were eligible to receive a combination therapy of sorafenib and transarterial chemoembolization. Enrollment took place from 3/2009 to 12/2011 at Johns Hopkins Hospital.
Pre-assignment Details: 90 patients consented and screened for study. 38 were ineligible and 2 later declined participation.
Groups:
- Sorafenib and Drug Eluting Beads: single arm
  sorafenib: sorafenib: given 400 mg twice per day for as long as it is beneficial
  LC Bead-TACE: LC Beads loaded with doxorubicin
  Doxorubicin loaded LC Beads: given intra-arterially into the liver, up to fours times in a 6 month period
Period: Overall Study
Arm/Group | Sorafenib and Drug Eluting Beads
Started (Patients evaluable for survival and safety analysis, and started on sorafenib) | 50
Patients Who Received TACE | 48 (2 patients withdrawn at Week 1 prior to TACE for intolerance to sorafenib)
Completed (Patients evaluable for time to progression analysis) | 46
Not Completed | 4
Not completed — Bridged to liver transplant | 3
Not completed — Bridged to resection | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib and Drug Eluting Beads
Number analyzed (Participants) | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [35 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 38
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Safety Will be Assessed by Grading Toxicities Reported at Intervals Throughout the Study. Higher Grade Toxicities Will be Assessed for Their Degree of Relatedness to the Study Treatment.
Description: Treatment toxicities assessed by CTCAE v3.0 were stratified by cycle - patients on Cycle 1, and patients on Cycles 2-5 or more. 50 patients were reviewed for toxicities for Cycle 1, and all 50 patients experienced at least one adverse event during this time period.
Time Frame: 6 weeks (Cycle 1)
Measure: Number; unit: # of participants with adverse events
Arm/Group | Sorafenib and Drug Eluting Beads
Number analyzed (Participants) | 50
# of participants with adverse events
  Anemia | 13
  Lymphopenia | 24
  Thrombocytopenia | 8
  Arrhythmia | 4
  Chest pain | 2
  Dissection | 1
  Embolus or coagulopathy | 1
  Hypertension | 7
  Lower extremity edema | 12
  Fatigue | 42
  Fever | 15
  Hand-foot skin reaction | 23
  Mucositis | 11
  Rash | 26
  Skin pain | 4
  Ascites | 3
  Anorexia | 28
  Diarrhea | 19
  Nausea or vomiting | 24
  Epistaxis or hemoptysis | 1
  Hematochezia | 2
  Hematoma | 3
  Tumor rupture | 1
  Elevated ALT level | 25
  Elevated AST level | 24
  Elevated AP level | 17
  Elevated amylase level | 10
  Elevated lipase level | 15
  Elevated INR level | 16
  Hyperbilirubinemia | 30
  Hypoalbuminemia | 27
  Infection | 6
  Dizziness | 4
  Headache | 9
  Encephalopathy | 3
  Nonspecific abdominal pain | 24
  Musculoskeletal pain | 24
  Right upper quadrant pain | 24
  Pain - other | 12
  Acute renal failure | 3
  Death (disease progression) | 1

2. Primary Outcome: Safety Will be Assessed by Grading Toxicities Reported at Intervals Throughout the Study. Higher Grade Toxicities Will be Assessed for Their Degree of Relatedness to the Study Treatment.
Description: Treatment toxicities assessed by CTCAE v3.0 were stratified by cycle - patients on Cycle 1, and patients on Cycles 2-5 or more.
Time Frame: 2 years (Cycles 2-5+)
Population: 39 patients were reviewed for toxicities for Cycle 2-5+. 11 patients out of the original 50 exited the study prior to Cycle 2.
Measure: Number; unit: # of participants with adverse events
Arm/Group | Sorafenib and Drug Eluting Beads
Number analyzed (Participants) | 39
# of participants with adverse events
  Anemia | 14
  Lymphopenia | 19
  Pancytopenia | 1
  Thrombocytopenia | 11
  Arrhythmia | 2
  Chest pain | 1
  Hypertension | 4
  Lower extremity edema | 3
  Fatigue | 30
  Fever | 4
  Hand-foot skin reaction | 20
  Mucositis | 6
  Rash | 12
  Skin pain | 3
  Ascites | 2
  Anorexia | 14
  Diarrhea | 15
  Nausea or vomiting | 13
  Epistaxis or hemoptysis | 1
  Cholangitis | 1
  Elevated ALT level | 9
  Elevated AST level | 10
  Elevated AP level | 15
  Elevated amylase level | 7
  Elevated lipase level | 9
  Elevated INR level | 8
  Hyperbilirubinemia | 11
  Hypoalbuminemia | 14
  Infection | 8
  Liver abscess | 1
  Dizziness | 1
  Headache | 6
  Encephalopathy | 3
  Nonspecific abdominal pain | 22
  Musculoskeletal pain | 17
  Right upper quadrant pain | 10
  Pain - other | 4
  Acute renal failure | 1
  Death (disease progression) | 2

3. Secondary Outcome: Efficacy Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) to Determine Response and Disease Control Rate
Description: Efficacy as assessed by radiographic tumor response using the RECIST criteria at baseline and at 6 months post the initiation of treatment. 33 out of the original 50 patients were evaluable at this time point, with 17 out of the 50 exiting prior to 6 months or were not assessable by RECIST criteria.
  Complete response (CR): Disappearance of all lesions targeted with therapy Partial Response (PR): at least 30% decrease in sum of longest diameter (LD) of targeted lesions Progressive Disease (PD): at least 20% increase in the sum of LD of targeted lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR or sufficient increase to qualify for PD
Time Frame: 6 months
Population: 33 out of the original 50 patients were evaluable for this outcome, with 17 out of the original 50 exiting prior to 6 months or were not assessable by RECIST criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib and Drug Eluting Beads
Number analyzed (Participants) | 33
Participants
  Complete Response | 1
  Partial Response or Stable Disease | 30
  Progressive Disease | 2
  Disease control rate (CR + PR + SD) | 31

4. Secondary Outcome: Efficacy Assessed by European Association for the Study of the Liver (EASL) Criteria to Determine Response and Disease Control Rate
Description: Efficacy as assessed by radiographic tumor response using the EASL criteria at baseline and at 6 months post the initiation of treatment.
  Complete response (CR): 100% tumor necrosis Partial Response (PR): more than 50% tumor necrosis Progressive Disease (PD): increase in tumor enhancement by more than 25% Stable Disease (SD): Cases that do not qualify for one of the above criteria
Time Frame: 6 months
Population: 32 out of the 50 patients had imaging assessable by EASL criteria at 6 months - 18 out of the original 50 had exited prior to this time point or did not have applicable imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib and Drug Eluting Beads
Number analyzed (Participants) | 32
Participants
  Complete Response | 7
  Partial Response | 15
  Stable Disease | 8
  Progressive Disease | 2
  Disease control rate (CR + PR + SD) | 30

5. Secondary Outcome: Efficacy - Median TTP After Combination Treatment With Sorafenib and TACE
Description: Time to progression (TTP) - defined as the time from initiation of therapy to disease progression (radiological). Median TTP calculated for all subjects and stratified by Barcelona Clinic Liver Cancer (BCLC) staging.
  46 patients out of 50 were reviewed for this outcome. 3 patients were excluded because they underwent liver transplantation and 1 patient was excluded for hepatic resection.
Time Frame: 3 years
Population: Median TTP stratified by BCLC staging; 3 patients had BCLC stage A disease, 14 with stage B, and 29 with stage C.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Sorafenib and Drug Eluting Beads
Number analyzed (Participants) | 46
months
  Median TTP | 13.9 [8.5 to 27.6]
  Median TTP for BCLC stage A: number analyzed (Participants) | 3
  Median TTP for BCLC stage A | 27.6 [15.8 to NA] — Number of patients insufficient to determine upper IQR
  Median TTP for BCLC stage B: number analyzed (Participants) | 14
  Median TTP for BCLC stage B | 24.7 [13.9 to 26.5]
  Median TTP for BCLC stage C: number analyzed (Participants) | 29
  Median TTP for BCLC stage C | 9.5 [5.2 to 12.8]

6. Secondary Outcome: Efficacy - Overall Survival (OS) After Combination Treatment With Sorafenib and TACE
Description: Overall survival was assessed with Kaplan-Meier estimates of survival, and the Mantel-Cox log-rank test was used to determine differences in survival.
  All 50 patients were included in survival analyses as all 50 received at least one dose of sorafenib.
Time Frame: 3 years
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Sorafenib and Drug Eluting Beads
Number analyzed (Participants) | 50
months | 20.4 [7.2 to 34.0]

7. Secondary Outcome: Efficacy - Factors Associated With Overall Survival (OS) After Combination Treatment With Sorafenib and TACE
Description: Overall survival was assessed with Kaplan-Meier estimates of survival, and the Mantel-Cox log-rank test was used to determine differences in survival.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: Hazard ratio
Arm/Group | Sorafenib and Drug Eluting Beads
Number analyzed (Participants) | 50
Hazard ratio
  Median liver tumor burden >10% | 2.60 [1.38 to 4.90]
  Median tumor size > 10cm | 2.12 [1.06 to 4.21]
  ECOG performance status | 2.45 [1.30 to 4.62]
  BCLC stage | 2.49 [1.39 to 4.44]

8. Other Pre Specified Outcome: Estimated Percentage of Participants Surviving After One Year
Description: Percentage of study patients surviving after one year from initial treatment analyzed with Kaplan-Meier curve.
Time Frame: 1 year
Population: All 50 patients were included in survival analyses as all 50 received at least one dose of sorafenib.
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib and Drug Eluting Beads
Number analyzed (Participants) | 50
percentage of participants | 64

9. Other Pre Specified Outcome: Estimated Percentage of Participants Surviving After Three Year
Description: Percentage of study patients surviving after three years from initial treatment analyzed with Kaplan-Meier curve.
Time Frame: 3 years
Population: All 50 patients were included in survival analyses as all 50 received at least one dose of sorafenib.
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib and Drug Eluting Beads
Number analyzed (Participants) | 50
percentage of participants | 19.6

10. Other Pre Specified Outcome: Median Overall Survival OS Stratified by BCLC Criteria
Description: Median overall survival stratified by Barcelona Clinic Liver Cancer (BCLC) staging as assessed by Kaplan-Meier estimator. Patients are grouped to stages A (early), B (intermediate), and C (advanced) according to stage of disease.
Time Frame: up to 4 years
Population: 50 total participants received sorafenib on trial. 3 were classified as BCLC A, 16 as BCLC B, and 31 as BCLC C.
Measure: Median (Full Range); unit: months
Arm/Group | Sorafenib and Drug Eluting Beads
Number analyzed (Participants) | 50
months
  BCLC A: number analyzed (Participants) | 3
  BCLC A | 45.6 [32.4 to 46.0]
  BCLC B: number analyzed (Participants) | 16
  BCLC B | 29.7 [12.1 to 34.5]
  BCLC C: number analyzed (Participants) | 31
  BCLC C | 8.0 [1.38 to 34.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the entire duration of study participation, an average of 2 years. Participants remained on study until further treatment with sorafenib and TACE was deemed to not be beneficial.
Arm/Group | Sorafenib and Drug Eluting Beads
All-Cause Mortality (participants affected / at risk) | 3/50
Serious Adverse Events (participants affected / at risk) | 8/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib and Drug Eluting Beads (N=50)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Elevated creatinine (Metabolism and nutrition disorders) | 1 (1)
Overdose on pain medication (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Tumor rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib and Drug Eluting Beads (N=50)
Anemia (Blood and lymphatic system disorders) | 14 (27)
Lymhopenia (Investigations) | 24 (43)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Investigations) | 11 (19)
Arrhythmia (Cardiac disorders) | 4 (4)
Non-cardiac chest pain (General disorders) | 1 (1)
Common hepatic artery dissection (Vascular disorders) | 1 (1)
Embolus or coagulopathy (Vascular disorders) | 1 (1)
Edema - lower extremity (General disorders) | 12 (15)
Fatigue (General disorders) | 42 (72)
Fever (General disorders) | 15 (19)
Hand foot skin reaction (Skin and subcutaneous tissue disorders) | 23 (43)
Mucositis (Gastrointestinal disorders) | 11 (17)
Rash (Skin and subcutaneous tissue disorders) | 26 (38)
Skin pain (Skin and subcutaneous tissue disorders) | 4 (7)
Ascites (Gastrointestinal disorders) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 28 (42)
Diarrhea (Gastrointestinal disorders) | 19 (34)
Nausea or vomiting (Gastrointestinal disorders) | 24 (37)
Epistaxis or hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hematochezia (Gastrointestinal disorders) | 2 (2)
Hematoma (Vascular disorders) | 3 (3)
Elevated ALT (Investigations) | 25 (34)
Elevated AST (Investigations) | 24 (34)
Elevated AP (Investigations) | 17 (32)
Elevated amylase (Investigations) | 10 (17)
Elevated lipase (Investigations) | 15 (24)
Elevated INR (Investigations) | 16 (24)
Hyperbilirubinemia (Investigations) | 30 (41)
Hypoalbuminemia (Investigations) | 27 (41)
Infection (Infections and infestations) | 8 (8)
Liver abscess (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 9 (15)
Encephalopathy (Nervous system disorders) | 2 (2)
Nonspecific abdominal pain (Gastrointestinal disorders) | 23 (45)
Pain - musculoskeletal (Musculoskeletal and connective tissue disorders) | 24 (41)
Pain - right upper quadrant (Gastrointestinal disorders) | 24 (34)
Pain - other (General disorders) | 12 (16)
Acute kidney injury (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes